CLINICAL TRIAL: NCT03283072
Title: Effects of Acute Intermittent Hypoxia on Sensory Function in Healthy Adults
Acronym: SensoryFLO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: IRB201700637
Record Dates: First submitted 2017-09-07; First posted 2017-09-14 (Actual); Results first posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Sensitivity
Keywords: thermal threshold; pressure pain threshold; temporal summation
MeSH Terms: conditions — Hypersensitivity

STUDY DESIGN:
Intervention Model Description: Within subjects design with randomization of presentation of four different hypoxia/normoxia intervals.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants can't see the device and therefore the settings. The assessment of sensory function is done by a separate investigator who did not participate in the set up of the hypoxicator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- Sequence 1 (Experimental): Intervention 1: 15 bouts of 2mins:1min hypoxia:hyperoxia Intervention 2: 15 bouts of 1mins:1min hypoxia:hyperoxia Intervention 3: 8 bouts of 2mins:1min hypoxia:hyperoxia 15 bouts of 1min:1min normoxia (sham)
  Interventions: Device: Intervention 1; Device: Intervention 2; Device: Intervention 3; Device: Intervention 4 (sham)
- Sequence 2 (Experimental): Intervention 2: 15 bouts of 1mins:1min hypoxia:hyperoxia Intervention 3: 8 bouts of 2mins:1min hypoxia:hyperoxia 15 bouts of 1min:1min normoxia (sham) Intervention 1: 15 bouts of 2mins:1min hypoxia:hyperoxia
  Interventions: Device: Intervention 1; Device: Intervention 2; Device: Intervention 3; Device: Intervention 4 (sham)
- Sequence 3 (Experimental): Intervention 3: 8 bouts of 2mins:1min hypoxia:hyperoxia 15 bouts of 1min:1min normoxia (sham) Intervention 1: 15 bouts of 2mins:1min hypoxia:hyperoxia Intervention 2: 15 bouts of 1mins:1min hypoxia:hyperoxia
  Interventions: Device: Intervention 1; Device: Intervention 2; Device: Intervention 3; Device: Intervention 4 (sham)
- Sequence 4 (Experimental): 15 bouts of 1min:1min normoxia (sham) Intervention 1: 15 bouts of 2mins:1min hypoxia:hyperoxia Intervention 2: 15 bouts of 1mins:1min hypoxia:hyperoxia Intervention 3: 8 bouts of 2mins:1min hypoxia:hyperoxia
  Interventions: Device: Intervention 1; Device: Intervention 2; Device: Intervention 3; Device: Intervention 4 (sham)

INTERVENTIONS:
Device: Intervention 1 — 15 bouts of 2mins:1min hypoxia:hyperoxia
Device: Intervention 2 — 15 bouts of 1mins:1min hypoxia:hyperoxia
Device: Intervention 3 — 8 bouts of 2mins:1min hypoxia:hyperoxia
Device: Intervention 4 (sham) — 15 bouts of 1min:1min normoxia

SUMMARY:
Exposure to acute intermittent hypoxia (AIH) can facilitate of motor output but no studies of sensory effects has been reported.

DETAILED DESCRIPTION:
Despite the strong results of motor studies, the affects of AIH on sensory function has not been established. We will use a commercially-available hypoxicator that can be programmed to achieve a targeted level of arterial oxygen saturation. We plan to compare 3 previously published protocols that have generated motor facilitation (and a sham condition) to characterize and effects on sensory function in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 40 years of age

Exclusion Criteria:

* Diagnosis of cardiovascular disease (Hypertension, arrhythmias, coronary artery disease, congenital and valvar heart diseases)
* Diagnosis of neuromuscular disease
* Diagnosis of any neurological disease
* Presence of concurrent medical illness including infection, fractures
* Diagnosis of obstructive sleep apnea
* Diagnosis of obstructive/restrictive lung disease
* Diagnosis of exercise induced asthma
* FEV1/FVC<80% and/or FVC<80% of predicted value indicating airway obstruction
* Subjects on prednisolone therapy or selective serotonin reuptake inhibitor (SSRI) therapy will be excluded from the study as these pharmacological agents are known to amplify the effects of IH[22, 23]
* Diagnosis of epilepsy or history of seizures and attention deficit disorders
* Pregnancy
* Diabetes
* History of coagulation disorders
* History of chronic pain
* Body mass index(BMI)> 35kg/m2
* Subjects on prescription medicines such as beta blockers and other drugs that are prescribed in any of the exclusionary disorders listed above.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2017-09-18 (Actual); Primary Completion 2020-07-06 (Actual); Study Completion 2020-07-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark D Bishop, PhD, Principal Investigator — University of Florida
Locations (1):
- Unversity of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Sequence 1: 1. 15 bouts of 2mins:1min hypoxia:hyperoxia
  2. 15 bouts of 1mins:1min hypoxia:hyperoxia
  3. 8 bouts of 2mins:1min hypoxia:hyperoxia
  4. 15 bouts of 1min:1min normoxia
- Sequence 2: 2. 15 bouts of 1mins:1min hypoxia:hyperoxia 3. 8 bouts of 2mins:1min hypoxia:hyperoxia 4. 15 bouts of 1min:1min normoxia
  1. 15 bouts of 2mins:1min hypoxia:hyperoxia
- Sequence 3: 3. 8 bouts of 2mins:1min hypoxia:hyperoxia 4. 15 bouts of 1min:1min normoxia
  1. 15 bouts of 2mins:1min hypoxia:hyperoxia
  2. 15 bouts of 1mins:1min hypoxia:hyperoxia
- Sequence 4: 4. 15 bouts of 1min:1min normoxia
  1. 15 bouts of 2mins:1min hypoxia:hyperoxia
  2. 15 bouts of 1mins:1min hypoxia:hyperoxia
  3. 8 bouts of 2mins:1min hypoxia:hyperoxia
Period: Overall Study
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4
Started | 7 | 5 | 5 | 5
Completed | 5 | 5 | 5 | 5
Not Completed | 2 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Sequence 1: 15 bouts of 2mins:1min hypoxia:hyperoxia 15 bouts of 1mins:1min hypoxia:hyperoxia 8 bouts of 2mins:1min hypoxia:hyperoxia 15 bouts of 1min:1min normoxia
- Sequence 2: 15 bouts of 1mins:1min hypoxia:hyperoxia 8 bouts of 2mins:1min hypoxia:hyperoxia 15 bouts of 1min:1min normoxia 15 bouts of 2mins:1min hypoxia:hyperoxia
- Sequence 3: 8 bouts of 2mins:1min hypoxia:hyperoxia 15 bouts of 1min:1min normoxia 15 bouts of 2mins:1min hypoxia:hyperoxia 15 bouts of 1mins:1min hypoxia:hyperoxia
- Sequence 4: 15 bouts of 1min:1min normoxia 15 bouts of 2mins:1min hypoxia:hyperoxia 15 bouts of 1mins:1min hypoxia:hyperoxia 8 bouts of 2mins:1min hypoxia:hyperoxia
- Total: Total of all reporting groups
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Total
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.4 (6.3) | 19.2 (1.1) | 20.8 (2.0) | 20.8 (2.1) | 22.0 (5.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 3 | 0 | 10
  Male | 1 | 2 | 2 | 5 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 3 | 2 | 1 | 3 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 2 | 3 | 3 | 1 | 9
  More than one race | 0 | 0 | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 5 | 5 | 5 | 20

OUTCOME MEASURES:

1. Primary Outcome: Sensory Function
Description: Thermal thresholds. Average reported.
Time Frame: Every 10 minutes for 60 minutes post intervention, average reported
Population: A 2-way analysis of co-variance with repeated measures (time*intervention) was conducted with gender as the covariate.
Measure: Mean (Standard Deviation); unit: Degrees celsius
Groups:
- Intervention 1: 1) 15 bouts of 1 minute hypoxia:1 minute hyperoxia;
- Intervention 2: 2) 15 bouts of hypoxia for 2 minutes, normoxia to hyperoxia 1 minute;
- Intervention 3: 3) 8 bouts of hypoxia for 2 minutes, normoxia to hyperoxia 1 minute;
- Intervention 4 (Sham): 4) normoxia
Arm/Group | Intervention 1 | Intervention 2 | Intervention 3 | Intervention 4 (Sham)
Number analyzed (Participants) | 20 | 20 | 20 | 20
Degrees celsius | 46.7 (1.5) | 46.4 (1.9) | 46.1 (1.9) | 45.9 (2.1)
Statistical Analysis 1: Comparison: Intervention 1 vs Intervention 2 vs Intervention 3 vs Intervention 4 (Sham); Test type: Superiority; p = 0.592, ANCOVA; Within, within repeated measures ANCOVA (gender as co-variate)

2. Primary Outcome: Temporal Sensory Summation
Description: Temporal summation represents increases in ratings of pain intensity measured using a numeric pain rating scale (0-no pain to 100-worst pain imaginable) to repeated heat stimuli of the same intensity; that is, "summation" represents increases in participant ratings of pain despite the maintenance of a standard temperature and is calculated as the difference between pain rating 1 and pain rating 6. Positive difference scores indicate that pain reported increased over the 6 pulses of heat. Here, the average difference across participants and over time is reported.
Time Frame: Every 10 minutes for 60 minutes post intervention, average reported
Population: 2-way repeated measures ANOVA with gender as the covariate
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Intervention 1: 15 bouts of 1 minute hypoxia:1 minute hyperoxia
- Intervention 2: 15 bouts of hypoxia for 2 minutes, normoxia to hyperoxia 1 minute
- Intervention 3: 8 bouts of hypoxia for 2 minutes, normoxia to hyperoxia 1 minute
- Intervention 4 (Sham): normoxia
Arm/Group | Intervention 1 | Intervention 2 | Intervention 3 | Intervention 4 (Sham)
Number analyzed (Participants) | 20 | 20 | 20 | 20
score on a scale | 17.4 (13.3) | 11.7 (10.2) | 10.9 (11.2) | 11.9 (15.6)
Statistical Analysis 1: Comparison: Intervention 1 vs Intervention 2 vs Intervention 3 vs Intervention 4 (Sham); Test type: Superiority; p = 0.721, ANCOVA; Within, within repeated measures ANCOVA (gender as co-variate)

3. Primary Outcome: Sensory Function - Pressure
Description: Pressure threshold is the force at which the sensation of pressure first is considered painful by the participant, average reported
Time Frame: Every 10 minutes for 60 minutes post intervention, average reported
Population: A 2-way analysis of co-variance with repeated measures (time*intervention) was conducted with gender as the covariate.
Measure: Mean (Standard Deviation); unit: kilograms force
Groups:
- Intervention 1: 1. 15 bouts of 2mins:1min hypoxia:hyperoxia
- Intervention 2: 2. 15 bouts of 1mins:1min hypoxia:hyperoxia
- Intervention 3: 3. 8 bouts of 2mins:1min hypoxia:hyperoxia
Arm/Group | Intervention 1 | Intervention 2 | Intervention 3 | Intervention 4 (Sham)
Number analyzed (Participants) | 20 | 20 | 20 | 20
kilograms force | 4.4 (3.4) | 4.6 (2.5) | 4.3 (2.8) | 4.3 (3.1)
Statistical Analysis 1: Comparison: Intervention 1 vs Intervention 2 vs Intervention 3 vs Intervention 4 (Sham); Test type: Superiority; p = 0.553, ANCOVA; Within, within repeated measures ANVOA (gender as covariate)

ADVERSE EVENTS:
Time Frame: 2 weeks
Description: The definitions do not differ
Groups:
- All Participants: All participants completed each protocol in a a randomly assigned order. Therefore all adverse event data are combined.
  1. 15 bouts of 2mins:1min hypoxia:hyperoxia
  2. 15 bouts of 1mins:1min hypoxia:hyperoxia
  3. 8 bouts of 2mins:1min hypoxia:hyperoxia
  4. 15 bouts of 1min:1min normoxia
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/22
Serious Adverse Events (participants affected / at risk) | 0/22
Other Adverse Events (participants affected / at risk) | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-18): https://cdn.clinicaltrials.gov/large-docs/72/NCT03283072/Prot_SAP_000.pdf